CLINICAL TRIAL: NCT06873295
Title: Evaluation of the Management Strategy for Acute Cholecystitis in the Digestive Surgery Department and Geriatric Intraoperative Unit in Subjects Over and Under 75 Years of Age
Brief Title: Management Strategy for Acute Cholecystitis in the Digestive Surgery Department and Geriatric Unit in Subjects Over and Under 75 Years
Acronym: GERBILLE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local /2023
Record Dates: First submitted 2023-06-22; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The management of these often frail elderly patients, with more comorbidities and declining functional capacities, is more complex and justifies a specific, tailored approach.

Age is also associated with an increasing prevalence of gallstones. The disadvantages of "cold" surgery (longer hospital stay, higher cost, risk of disease recurrence in the interim, difficult surgery with more scar tissue due to repeated inflammation) have to be weighed against the high operative risk in the case of emergency surgery, leading to strict criteria for early cholecystectomy.

These criteria are rarely met in geriatric patients, who thus enter a hospital cycle whose impact on morbidity and mortality, as well as on loss of autonomy, has been demonstrated in this population. What's more, the deteriorating general condition of frail elderly patients means that a number of them end up being definitively rejected for surgery, despite an initial strategy of cold cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Diagnosis of acute cholecystitis.
* Hospitalization in the digestive surgery department and geriatric perioperative unit of Nîmes University Hospital.

Exclusion Criteria:

* Patients under 18 years of age.
* Opposition of the patient to his inclusion in the study after sending the letter of information and non-opposition.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the digestive surgery department and geriatric perioperative unit of the CHU de Nîmes with a diagnosis of acute cholecystitis.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Rate of patients with an initial cold cholecystectomy strategy who did not undergo surgery, died or underwent emergency surgery | Up to 6 months, from date of first collection to date of end of collection
  Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Simonet Anne Clarisse, Nîmes, France